

# **Statistical Analysis Plan**

| Protocol Title: | Multicenter, Safety and Efficacy, Open-Label Extension Study of ACTIMMUNE® (interferon γ-1b) in Children and Young Adults with Friedreich's Ataxia |
|---|---|
| Protocol Number: | HZNP-ACT-302 Version 2.0 Amendment 1 (28-SEP-2016) |
| Compound: | ACTIMMUNE |
| Phase: | III |
| Sponsor: | Horizon Pharma Ireland Ltd. Connaught House, 1 <sup>st</sup> Floor 1 Burlington Road Dublin 4, Ireland |
| SAP Author: | Premier Research Group Limited<br>387 Shuman Boulevard, STE 340W<br>Naperville, IL, 60563 |
| SAP Version: | Final Version 1.0 |
| SAP Date: | 22-MAY-2017 |

CONFIDENTIAL

Final Version 1.0

# **DOCUMENT HISTORY**

| Version | Date | Author | Description |
|---|---|---|---|
| 0.1 | 14-OCT-2016 | | Initial Draft |
| 0.2 | 23-NOV-2016 | | Updated sponsor comments from original draft |
| 0.3 | 09-MAY-2017 | | <ul> <li>Updated to keep only Safety population,</li> <li>Tables will only have overall column,</li> <li>Remove all efficacy analyses,</li> <li>Analysis from Baseline of HZNP-ACT-301 to Week 26 of HZNP-ACT-302 (52-week treatment duration) will not be performed</li> <li>Updated TOC to reflect removed analyses,</li> <li>added note that analyses is only for abbreviated CSR report</li> </ul> |
| 1.0 | 22-MAY-2017 | | Updated for finalization of Document |

# SIGNATURE PAGE AND APPROVALS



Protocol: HZNP-ACT-302


# TABLE OF CONTENTS

| DO | CUMEN | NT HISTORY | 2 |
|-----------|--------|-------------------------------------------------|----|
| SIG | NATUF | RE PAGE AND APPROVALS | 3 |
| TAE | BLE OF | CONTENTS | 4 |
| ABE | BREVIA | ATIONS | 6 |
| 1. | OVE | ERVIEW | 7 |
| 2. | STU | DY OBJECTIVES AND ENDPOINTS | 7 |
| | 2.1 | Study Objectives | 7 |
| | | 2.1.1 Primary Objective | 7 |
| | | 2.1.2 Secondary Objectives | 8 |
| | 2.2 | Study Endpoints | 8 |
| | | 2.2.1 Safety Endpoints | 8 |
| 3. | OVE | ERALL STUDY DESIGN AND PLAN | 8 |
| 4. | ANA | ALYSIS AND REPORTING | 12 |
| | 4.1 | Interim Analysis | 12 |
| | 4.2 | Final Analysis | 12 |
| <b>5.</b> | ANA | ALYSIS POPULATIONS | 12 |
| | 5.1 | Sample Size | 12 |
| 6. | GEN | NERAL ISSUES FOR STATISTICAL ANALYSIS | 12 |
| | 6.1 | Visit Windows | 13 |
| | 6.2 | Data Adjustments, Handling, Conventions | 13 |
| | 6.3 | Derived and Computed Variables | 13 |
| <b>7.</b> | STU | DY SUBJECTS AND DEMOGRAPHICS | 14 |
| | 7.1 | Disposition of Subjects and Withdrawals | 14 |
| | 7.2 | Protocol Violations and Deviations | 14 |
| | 7.3 | Demographics and Other Baseline Characteristics | 14 |
| 8. | EFF | ICACY ANALYSIS | 15 |
| 9. | SAF | ETY AND TOLERABILITY ANALYSIS | 15 |
| | 9.1 | Adverse Events | 16 |
| | | 9.1.1 Deaths | 16 |
| | 9.2 | Clinical Laboratory Evaluations | 16 |
| | | 9.2.1 Immunogenicity Testing | 16 |
| | 9.3 | Vital Signs | 16 |

| | 9.4 | Electrocardiogram (ECG) and Echocardiogram | 17 |
|-----|-----|--------------------------------------------|----|
| | 9.5 | Concomitant Medication | 17 |
| | 9.6 | Exposure and Compliance | 17 |
| 10. | CHA | ANGES FROM PLANNED ANALYSIS | 17 |
| 11. | REF | ERENCES | 17 |
| 12. | TAB | BLES, LISTINGS, AND FIGURES | 18 |
| 13. | PLA | NNED TABLES | 20 |
| 14. | PLA | NNED LISTINGS | 21 |

Protocol: HZNP-ACT-302 


# **ABBREVIATIONS**

| ABBREVIATION | DEFINITION OR DESCRIPTION |
|---|---|
| 9-HPT | 9-hole peg test |
| ADA | Anti-Drug Antibody |
| ADL | Activities of Daily Living |
| AE | Adverse Event |
| ATC | Anatomical Therapeutic Chemical |
| BSA | Body Surface Area |
| CI | Confidence Interval |
| CRF | Case Report Form |
| DSMB | Data Safety Monitoring Board |
| CSR | Clinical Study Report |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| FA | Friedreich's Ataxia |
| FARS | Friedreich's Ataxia Rating Scale |
| FARS-mNeuro | Friedreich's Ataxia Rating Scale excluding the peripheral nervous system |
| | subscale score and the facial and tongue atrophy and fasciculations from |
| | the bulbar subscale score |
| FARStot | Total FARS Score |
| FDA | Food and Drug Administration |
| ICH | International Conference on Harmonisation |
| IFN | interferon |
| LCSLC | Low-contrast sloan letter chart |
| LLOQ | Lower Limit of Quantitation |
| LOD | Limit of Detection |
| LiSN-S | Listening in Spatialized Noise-Sentences Auditory Test |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MFIS | Modified Fatigue Impact Score |
| NAb | Neutralizing Antibody |
| PedsQL | Pediatric Quality of Life |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SF-36 | 36-item short-form health survey |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| T25FW | Timed 25-foot-walk |
| TIW | Three times a week |
| TEAE | Treatment-emergent Adverse Event |
| ULOQ | Upper Limit of Quantitation |
| WHO-DD | World Health Organization Drug Dictionary |

Protocol: HZNP-ACT-302 


#### 1. OVERVIEW

This Statistical Analysis Plan (SAP) describes the planned analysis and reporting for Horizon Pharma Ireland, Ltd. protocol HZNP-ACT-302 (Multicenter, Safety and Efficacy, Open-Label Extension Study of ACTIMMUNE® (interferon γ-1b) in Children and Young Adults with Friedreich's Ataxia), Final Version 2.0 incorporating Amendment 1, dated 28-SEP-2016.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials [1]. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association [2] and the Royal Statistical Society [3], for statistical practice.

The planned analysis identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analysis not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc, or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

In addition to the study protocol, the following documents were reviewed in preparation of this SAP:

- The electronic case report forms (eCRFs) for this Protocol
- ICH Guidance on Statistical Principles for Clinical Trials (E9).

The reader of this SAP is encouraged to also read the clinical protocol, and other identified documents, for details on the planned conduct of this study. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

#### 2. STUDY OBJECTIVES AND ENDPOINTS

# 2.1 Study Objectives

# 2.1.1 Primary Objective

The primary objectives of this study are:

- To evaluate the long-term safety of ACTIMMUNE in subjects with Friedreich's Ataxia (FA).
- To evaluate the effect of ACTIMMUNE (interferon [IFN]-γ 1b) on the change from Baseline of HZNP-ACT-302 to Week 26 for all subjects and from Baseline of HZNP-ACT-301 to Week 26 of HZNP-ACT-302 (52-week treatment duration) for subjects receiving active treatment in both studies in neurological outcomes as measured by Friedreich's Ataxia Rating Scale (FARS) excluding the peripheral nervous system subscale score and the facial and tongue atrophy and fasciculations from the bulbar subscale score (FARS-mNeuro score).

Protocol: HZNP-ACT-302 


# 2.1.2 Secondary Objectives

The secondary objectives of this study are to evaluate the effect of ACTIMMUNE (interferon [IFN]-γ 1b) on the change from Baseline(HZNP-ACT-302) to Week 26 for all subjects and from Baseline of HZNP-ACT-301 to Week 26 of HZNP-ACT-302 (52-week treatment duration) for subjects receiving active treatment in both studies for the following:

- Activities of Daily Living (ADL)
- The timed 25-foot-walk-test (T25FW)
- Responder rate (≥3 point improvement in the FARS-mNeuro score)
- Neurological outcome as measured by the total FARS score (FARStot)

# 2.2 Study Endpoints

The analysis for this study is for an abbreviated safety Clinical Study Report (CSR). All efficacy endpoints mentioned in the protocol have been removed and noted as changes to the planned analyses.

# 2.2.1 Safety Endpoints

Adverse event and concomitant medication data will be summarized. Clinical laboratory safety data, vital sign data, echocardiogram data, and ECG interval data will be summarized with descriptive statistics for Baseline of HZNP-ACT-302, post-dose, and change from Baseline of HZNP-ACT-302 to post-dose values. Shift tables will be presented for clinical laboratory values and ECG categorical results from Baseline of HZNP-ACT-302 to each post-dose visit. Physical examination findings will be listed by subject. Results of immunogenicity testing will be presented in tabular format.

#### 3. OVERALL STUDY DESIGN AND PLAN

This is a multi-center, dose-escalation, open-label extension study of HZNP-ACT-301 examining the safety and efficacy of ACTIMMUNE in the treatment of FA in children and young adults. Subjects who complete 26 weeks of blinded treatment in HZNP-ACT-301 will be eligible for enrollment in this study. In order to maintain the study blind in HZNP-ACT-301, all subjects in the open-label extension study will undergo ACTIMMUNE titration, regardless of treatment received in HZNP-ACT-301. The sample size is not based on statistical considerations.

The overall maximum treatment duration for an individual subject is expected to be 26 weeks, with a Follow-Up Safety Visit two weeks following last dose of study drug. As per the study design and schedule of events below (Table 1, Table 2), subjects will all be assigned to start on ACTIMMUNE 10  $\mu$ g/m² in the first week. This will be followed by weekly escalation to 25, 50, and 100  $\mu$ g/m²three times a week (TIW) on Days 8, 15, and 22, respectively. The study drug dose is planned to be escalated on a weekly basis over the first 4 weeks of treatment (from  $10\mu$ g/m²to 100  $\mu$ g/m²), however, the dose may be reduced, interrupted, or held based on tolerability. By Week 13, all subjects are to be on a stable tolerated dose of study drug in order to continue study participation.

Protocol: HZNP-ACT-302 


Table 1. Study Design

# Schematic of Study Design



Week 26 of HZNP-ACT-301 will serve as the Baseline Visit (Day 1) for this study. Subjects will receive the last dose of the randomized drug from HZNP-ACT-301in a double-blind fashion, and the first dose of study drug for the open-label extension study (10 μg/m²) will be distributed for administration at home according to the planned TIW dosing schedule.

The planned dose escalation consists of two doses of ACTIMMUNE 10  $\mu$ g/m<sup>2</sup> in the first week, followed by weekly escalation to 25, 50, and 100  $\mu$ g/m<sup>2</sup> TIW on Days 8, 15, and 22, respectively; however, the dose may be reduced, interrupted, or held based on tolerability. All subjects are

to be on a stable tolerated dose of study drug by Week 13 in order to continue study participation.

Subjects and/or caregivers will be contacted by email or phone to monitor safety and dosing logistics on a weekly basis from Day 1 (Week 26 of HZNP-ACT-301) through Week 4 (or until stable tolerated dose is achieved) and on a monthly basis after Week 4 (or after dose stabilization) through Week 26.

Protocol: HZNP-ACT-302 


**Table 2.Schedule of Events** 

| Study Phase | Treatment Period | | | Follow-up | |
|---|---|---|---|---|---|
| Visit # | Baseline <sup>1</sup> | 1 2 3 | | | Safety Visit |
| Week | 1 | 4 | 13 | 26 (or PW) | 28 |
| Study Days (± visit window) | Day 1<br>(Week 26 of Study<br>HZNP-ACT-301) | 29 (± 3)<br>days | 92 (± 3)<br>days | 183 (± 3)<br>days | 197 (± 3)<br>days |
| Informed consent/assent | X | | | 1 | |
| Review of inclusion/exclusion criteria | X | | | | |
| Weight/height, BSA <sup>2</sup> | X | X | X | X | |
| Educate on dosing technique and schedule <sup>3</sup> | X | X | X | | |
| Dose given at study visit <sup>4</sup> | | X | X | X | |
| Dispense study drug | X | X | X | | |
| Drug compliance | | X | X | X | |
| Phone (email) contact for safety and dosing logistics <sup>6</sup> | X | X | X | | |
| Efficacy assessments <sup>7</sup> | | | | | |
| Functional staging of FA | X | | X | X | |
| FARS <sup>7</sup> | X | | X | X | |
| T25FW <sup>7</sup> | X | | X | X | |
| 9-HPT <sup>7</sup> | X | | X | X | |
| Vision testing (LCSLC) | X | | | X | |
| Auditory testing (LiSN-S) <sup>8</sup> | X | | | X | |
| Frataxin protein: whole blood, muscle biopsy (optional) <sup>9</sup> , and buccal cells | X | | X | X | |
| Physician and Patient Global assessments | X | | X | x | |
| ADL | X | | X | X | |
| Quality of Life (QOL) Assessments | | | | | |
| PedsQL or SF-36 <sup>10</sup> | X | | X | X | |
| MFIS | X | | X | X | |
| Safety Assessments | | | | | |
| TEAE, SAE assessment <sup>11</sup> | X | X | X | X | X |
| Immunogenicity testing <sup>12</sup> | X | X | X | X | X |
| Echocardiogram | X | | | X | |
| ECG | X | | X | X | |
| Physical examination <sup>13</sup> | X | X <sup>13</sup> | X | X | X <sup>13</sup> |
| Vital Signs: blood pressure, pulse, temperature | X | X | X | X | |
| Urine pregnancy test 14 | X | X | X | X | |
| Prior/concomitant medications | X | X | X | X | X |
| Clinical laboratory evaluation <sup>15</sup> | X | X | X | X | |
| (hematology, chemistry, urinalysis) | | | | | |
| End treatment | | | 1 | X | |
| O UPT-O belegant ADI posticities of Joily living DCA | | | | | |

9-HPT=9-hole peg test, ADL=activities of daily living, BSA=body surface area, ECG=electrocardiogram, FA=Friedreich's Ataxia, FARS=Friedreich's Ataxia Rating Scale, IFN=interferon, LCSLC=Low-contrast Sloan letter chart, LiSN-S=Listening in Spatialized Noise-Sentences Auditory Test, MFIS=Modified Fatique Impact Scale, PedsQL=Pediatric Quality of Life, PW=premature withdrawal, QOL=quality of life, SAE=serious adverse event, SF-36=36-item short form health survey, T25FW=timed 25-foot walk, TEAE=treatment-emergent adverse event.

Footnotes are presented on the next page.

Protocol: HZNP-ACT-302 


On Day 1 (Baseline), subjects will receive the last dose of assigned study drug (ACTIMMUNE or placebo) for HZNP-ACT-301, and undergo assessments; these assessments will serve as the Week 26 assessments for HZNP-ACT-301 and the Baseline assessments for HZNP-ACT-302.

Height and weight will be measured at Baseline/Day 1 (Week 26 of Study HZNP-ACT-301), and Weeks 4, 13, and 26 to determine BSA; dosing will be based on BSA at Baseline/Day1, and Weeks 4 and 13.

- Study drug will be initiated at home following the Baseline/Day 1 visit at 10 µg/m² according to the subject's TIW dosing schedule. The planned dose escalation consists of two doses of ACTIMMUNE 10 µg/m² in the first week, followed by weekly escalation to 25, 50, and 100 µg/m² TIW on Days 8, 15, and 22, respectively; however, the dose may be reduced, interrupted, or held based on tolerability. All subjects are to be on a stable tolerated dose of study drug by Week 13 in order to continue study participation
- At the Baseline/Day 1 visit (Week 26 of Study HZNP-ACT-301), subjects will receive the last dose of study drug from the double-blind Study HZNP-ACT-301 (ACTIMMUNE or placebo). The first dose for this open-label extension study (ACTIMMUNE 10µg/m²) will be administered at home before bedtime according to the subject's TIW dosing schedule. Dosing at Weeks 4, 13, and 26 will be performed at the clinic. All other doses will be administered at home before bedtime.
- Subjects will be given a 4-week supply of study drug prior to clinic discharge at the Baseline/Day 1 Visit (Week 26 of Study HZNP-ACT-301). At the Week 4 and 13 Visits, subjects will be given a 6-week supply of study drug, and additional study drug will be directly shipped to the subjects' homes as needed; if direct shipment is not feasible, subjects may receive a full supply at Weeks 4 and 13 (9-week supply at Week 4 and 13-week supply at Week 13).
- Subjects and/or caregivers will be contacted by email or phone to monitor safety and dosing logistics on a weekly basis during the dose-escalation period (from Day 1 through at least Week 4 [or later until a stable tolerated dose is reached]) and on a monthly basis after dose stabilization (from Week 4 or when dose is stabilized) through Week 26.
- Functional staging, FARS, T25W, and 9-HPT will be performed at approximately the same time of day at each visit and by the same examiner.
- The LiSN-S will only be performed for subjects who had a normal audiogram prior to enrollment in HZNP-ACT-301. The LiSN-S will be performed at the Baseline/Day 1 (Week 26 of Study HZNP-ACT-301) and Week 26 visits.
- Muscle biopsies will be optional for each subject, and consent will be signed prior to biopsy collection. Biopsies will be the last efficacy assessment of the day at Weeks 13 and 26.
- The PedsQL (study subject and parent/caregiver assessments) will be administered throughout the study for subjects who received the PedsQL at their Baseline Visit of the HZNP-ACT-301 study (even if subjects turn 18 during their participation in either Study HZNP-ACT-301 or HZNP-ACT-302). The SF-36 will continue to be administered throughout the study for subjects who completed the SF-36 during their HZNP-ACT-301 study participation.
- Adverse events occurring or worsening on or after the date of administration of the first dose of study drug at home through the end of the study will be considered treatment-emergent adverse events (TEAEs). All SAEs that occur on or after the date of administration of the first dose of study drug at home through two weeks after study discontinuation will be recorded.
- If a subject tests positive for anti-drug antibodies (ADA), he/she will be followed until ADA levels revert to baseline.
- Brief physical examinations will be performed at the Week 4 and Follow-Up Safety Visits; all other examinations will be complete physical examinations.
- <sup>14</sup> Only for female subjects of childbearing potential.
- 15 Collect blood samples for clinical safety laboratory testing (9.3 mL; 1.0 mL for hematology, 3.5 mL for chemistry, 3.0 mL discard, and 1.8 mL for PT/INR/aPTT) and a urine sample for urinalysis.

Protocol: HZNP-ACT-302 


#### 4. ANALYSIS AND REPORTING

# 4.1 Interim Analysis

No formal interim analysis is planned for this study, but the study will be monitored by a Data Safety Monitoring Board (DSMB), which will advise the Sponsor regarding the continuing safety of study subjects and potential subjects as well as the continuing validity and scientific merit of the trial.

# 4.2 Final Analysis

All final, planned analysis identified in the protocol and in this SAP will be performed after the last subject has completed the Follow-up Safety Visit and all relevant study data have been processed and integrated into the analysis data base.

Any post-hoc, exploratory analysis completed to support planned study analysis, which were not identified in this SAP, will be documented and reported in appendices to the CSR. Any results from these unplanned analyses (post-hoc) will also be clearly identified in the text of the CSR.

#### 5. ANALYSIS POPULATIONS

The following analysis populations are planned for this study:

• Safety Population (SAFETY): The Safety Population includes all subjects who receive at least one dose of open-label study drug after the Baseline Visit for HZNP-ACT-302. All analyses will be based on the Safety Population unless otherwise noted.

# 5.1 Sample Size

Subjects who complete 26 weeks of blinded treatment in Study HZNP-ACT-301 will be eligible for enrollment. The sample size is not based on statistical considerations; therefore no inference will be drawn from any statistical tests conducted.

#### 6. GENERAL ISSUES FOR STATISTICAL ANALYSIS

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed using SAS® Software (release 9.3 or higher) for Windows, unless otherwise specified.

Continuous (quantitative) variables will be summarized using descriptive statistics including number of non-missing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical (qualitative) variables will be summarized using the number and proportion of each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment group.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the raw data. Measures of location (mean and median) will be reported to 1 degree of precision more than the raw data and measures of spread (standard deviation) will be reported to two degrees of precision more than the raw data.

Assessments done on unscheduled visits will not be summarized but will be listed. All analyses will be completed on the Safety Population unless otherwise specified. Additionally, all summaries will be presented by overall treatment.

Protocol: HZNP-ACT-302 


All final, planned analyses identified in the protocol and in this SAP will be performed after all relevant study data have been processed and integrated into the analysis database, analysis populations have been finalized, and the database has been locked. Any post-hoc, exploratory analysis completed to support planned study analyses, which were not identified in this SAP, will be documented and reported in Section 9.8 of the CSR. Any results from these unplanned analyses (post-hoc) will also be clearly identified as subject in the text of the CSR.

#### **6.1 Visit Windows**

Subjects who withdraw from the study will have their data collected at the premature withdrawal (PW) visit assigned to the closest scheduled visit (either prior or post PW) where the data was scheduled to have been collected based on the protocol schedule of events. The data collected closest in time and date to protocol scheduled timing will be used for analysis.

# 6.2 Data Adjustments, Handling, Conventions

All collected data will be presented in listings. Data not subject to analyses according to this plan will not appear in any tables or graphics but will be included only in the data listings.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) (version 16.1). Concomitant medications will be coded using World Health Organization Drug Dictionary (WHO-DD) (version March 1, 2013).

If partial dates occur, the convention for replacing missing dates for the purposes of calculating derived variables is as follows:

If an AE has a missing severity, it will be imputed as 'Severe'; any missing relationship to study drug of an AE will be imputed as 'Related'. No other missing data will be imputed unless otherwise specified.

In general, for quantitative laboratory values reported as '<' or '≤', the lower limit of quantitation (LLOQ), or limit of detection (LOD), the reported value (i.e., LLOQ, LOD) will be used for analysis).

For quantitative laboratory values reported as '>' or '\geq', the upper limit of quantitation (ULOQ), the reported value (i.e., ULOQ) will be used for analysis.

For analysis purposes, repeat laboratory test results will not be used unless the original laboratory value is missing or indicated as invalid, in which case the first non-missing repeat laboratory value will be used for data analysis.

# **6.3** Derived and Computed Variables

The following derived and computed variables have been initially identified as important for the analyses of Safety, Efficacy and Exploratory endpoints. It is expected that additional variables may be required. The SAP will not be amended for additional variables that are not related to the primary target or key secondary target variables. Any additional derived or computed variables will be identified and documented in the SAS programs that create the analysis files. If the SAP is not amended, further derivations related to primary and secondary target variables will be described in the CSR.

• 302 Baseline = The last non-missing measurement/assessment on the date of Week 26 Visit from HZNP-ACT-301. If this measurement is missing or otherwise unavailable, it will be the last non-missing measurement/assessment on or prior to first dose in HZNP-

Protocol: HZNP-ACT-302 


ACT-302.

• 301 Baseline = The last non-missing measurement/assessment prior to first dose of Study in HZNP-ACT-301.

- Study Day = Assessment Date Date of Enrollment + 1
- Change from Baseline = Value at Post-Baseline Value at Baseline
- Concomitant Medication is defined as any medication a subject has received concurrently with study treatment.
- Prior Medication is defined as any medication or therapies initiated prior to date of first dose of study drug. Medications that are started prior to the date of first dose of study drug and continue after the first dose of drug are considered to be both prior and concomitant medications.
- Treatment-Emergent Adverse Event (TEAE) A TEAE is any adverse change from the subject's baseline condition that occurs on or after the date of the first dose of study drug through the duration of the clinical study.
- Related TEAE Any TEAE with a reported relationship to study drug of 'possibly related'.
- Compliance = Calculated as the percentage of the number of vials used divided by the expected number of vials used, where the number of vials used is the number of used vials returned.

#### 7. STUDY SUBJECTS AND DEMOGRAPHICS

# 7.1 Disposition of Subjects and Withdrawals

All subjects who provide informed consent/assent will be accounted for in this study. The number of subjects enrolled, completing, and withdrawing from the study, as well as reason for withdrawal, will be summarized by overall treatment. All disposition information will be included in a listing.

#### 7.2 Protocol Violations and Deviations

Protocol deviations will be collected by the clinical team and provided to Premier biostatistics prior to database lock. Deviations will be reviewed on a case-by-case basis to be classified as major or minor by the project team prior to database lock. Major and minor deviations will be included in a listing.

### 7.3 Demographics and Other Baseline Characteristics

Descriptive summaries and frequencies/percentages of demographic and other baseline characteristics will be completed for all enrolled subjects in the safety population for data collected in HZNP-ACT-301. These tabulations will include the following variables:

• Demographics (age, age categories (10-16 inclusive, and 17 and above), gender, race, ethnicity, height, weight, and Body Surface Area (BSA))

Tabulations of baseline HZNP-ACT-301 efficacy assessments will include the following in a separate table:

Protocol: HZNP-ACT-302 


- FA Functional Stage
- FARS-mNeuro score
- ADL
- T25FW
- FARStot

Descriptive summaries and frequencies/percentages of demographic and other baseline conditions in separate tabulations will include the following:

- Medical History
- Prior Medications
- Baseline Physical Examination

Medical History: Incidences of findings in medical history will be summarized by System Organ Class and preferred term.

Prior Medications: The frequency and percentage of all prior medications will be summarized by Anatomical Therapeutic Chemical (ATC) classifications level 3 and preferred term for all subjects. Subjects will only be counted once within ATC and preferred term. These data will be grouped by overall treatment.

Baseline physical examination: Baseline physical examination will be summarized by body system and result by overall treatment.

#### 8. EFFICACY ANALYSIS

All analyses are being conducted for an abbreviated safety CSR, and no efficacy analysis will be carried out.

# 9. SAFETY AND TOLERABILITY ANALYSIS

The analysis of safety assessments in this study will include summaries of the following categories of safety and tolerability data collected for each subject:

- Adverse Events
  - o Summary of all Adverse Events
  - o TEAEs, and Serious Adverse Events (SAEs)
  - o TEAEs by severity
  - o TEAEs by relationship to study drug
  - o TEAEs leading to premature withdrawal
  - o Any deaths
- Clinical Laboratory Investigations
  - o Complete Blood Count
  - o PT, INR, and aPTT
  - o Chemistry panel
  - Urinalysis
  - Immunogenicity samples
- Electrocardiograms (ECG)
- Echocardiograms
- Physical Examinations
- Concomitant Medications

Protocol: HZNP-ACT-302 


• Study Drug Exposure and Treatment Compliance

All tabulations and summaries for these categories will be performed on the safety population unless otherwise noted.

#### 9.1 Adverse Events

Missing and partially missing AE start and/or stop dates will be imputed for the purpose of statistical analysis, according to the specifications described in Section 6.1.

A summary of overall TEAEs, TEAEs, SAEs, TEAEs leading to PW, TEAEs by relationship to study drug, and severity of TEAEs will be presented by overall treatment.

Summaries and incidence rates (frequencies and percentages) of individual TEAEs by MedDRA System Organ Class (SOC) and preferred term will be displayed by overall treatment received. Such summaries will be displayed for TEAEs, SAEs, TEAEs leading to early termination, TEAEs by relationship to study drug, and TEAEs by severity

Each subject will be counted only once within each preferred term. If a subject experiences more than one TEAE within a preferred term only the TEAE with the strongest relationship or the maximum intensity, as appropriate, will be included in the summaries of relationship and intensity. No inferential statistical tests will be performed.

In the AE data listings, all AEs will be displayed. AEs that are not treatment-emergent will be flagged.

#### 9.1.1 Deaths

A summary and data listing of deaths that occurred will be provided, displaying details of the event(s) captured on the CRF.

#### 9.2 Clinical Laboratory Evaluations

Descriptive summaries of actual (absolute) values and changes from baseline will be presented for Chemistry, Urinalysis, Complete Blood Count, PR, INR, and aPTT. These tables will be grouped by visit, and overall treatment.

The number and proportion of subjects with clinical laboratory values below, within, or above normal ranges, at each study visit will be tabulated (shift tables) for each clinical laboratory analyte by treatment group. Normal ranges will be provided by the central laboratory (URMC) used in this study.

Laboratory values will be displayed in data listings and those that are outside the normal range will be flagged, along with the corresponding normal ranges.

# 9.2.1 Immunogenicity Testing

Frequency and percentages of positive anti-drug antibodies (ADA) and neutralizing antibodies (NAb) will be summarized by scheduled visit, and overall treatment received. Additionally, immunogenicity data will be presented in a data listing.

# 9.3 Vital Signs

Descriptive summaries of actual (absolute) values and changes from baseline will be presented for all vital signs (temperature, systolic blood pressure, diastolic blood pressure, heart rate),

Protocol: HZNP-ACT-302 


weight, height, and BSA will be presented by visit and overall treatment. These data will be presented in a data listing by subject.

# 9.4 Electrocardiogram (ECG) and Echocardiogram

Descriptive summaries of actual (absolute) values and changes from baseline will be presented for ECG quantitative measures (heart rate, PR interval, QRS duration, QT interval and QTC interval). These data will be summarized by visit and overall treatment.

Additionally, the frequency and percentage of subjects with normal, abnormal not clinically significant, and abnormal clinically significant ECGs will be summarized by visit. Shift tables will also be presented and display the number of subjects who had values that shifted from their baseline result.

Echocardiogram data will be summarized for left ventricular hypertrophy, left ventricle dilated, ejection fraction (%), PWTd (cm), IVSTd (cm), LVOT peak velocity (m/sec), LVOT obstruction (y/n).

Left centricular hypertrophy, left ventricle dilated and LVOT obstruction will be counted by the frequency and percentage of subjects with, without, and unknown within ventricular category. Ejection fraction, PWTd (cm), IVSTd (cm), and LVOT peak velocity (m/sec), will be summarized by descriptive statistics.

ECG and Echocardiogram data will be presented by subject in separate data listings.

#### 9.5 Concomitant Medication

Concomitant medications will be analyzed the same way as prior medications as noted in Section 7.3. The frequency and percentage of all concomitant medications will be summarized by ATC classification level 3 and preferred term for all subjects. Subjects will only be counted once within ATC and preferred term. These data will be grouped by overall treatment. A listing of prior and concomitant medications will be presented by subject.

#### 9.6 Exposure and Compliance

For each subject, treatment compliance and exposure will be calculated and summarized for the entire study. Overall compliance and exposure will be summarized and grouped by overall treatment. Compliance is defined in Section 6.3. Drug accountability, exposure, and treatment compliance will also be provided in a subject listing.

# 10. CHANGES FROM PLANNED ANALYSIS

All efficacy analyses has been removed from the study as described in the protocol.

#### 11. REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.

ASA. (1999) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, August 7, 1999. <a href="http://www.amstat.org/about/ethicalguidelines.cfm">http://www.amstat.org/about/ethicalguidelines.cfm</a>

RSS. (1993) The Royal Statistical Society: Code of Conduct, April 1993. http://www.rss.org.uk/main.asp?page=1875.

Protocol: HZNP-ACT-302 


#### 12. TABLES, LISTINGS, AND FIGURES

This section presents the list of shells for the planned Tables, Listings and Figures to be programmed in support of the planned analyses identified in the SAP. This section is intended to support the SAP and provides guidance on the programming specifications (shells) for the planned outputs and may be updated, independent of the SAP, with any updates appropriately documented, reviewed, and approved.

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

# **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, superscripted and subscripted text will not be used in tables and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing. Hexadecimal character representations are allowed (e.g.,  $\mu$ ,  $\alpha$ ,  $\beta$ ).
- All titles will be centered on a page. The ICH numbering convention is to be used for all outputs.
- All footnotes will be left justified and at the bottom of a page.
- Missing values for both numeric and character variables will be presented as blanks in a table or data listing. A value of zero may be used if appropriate to identify when the frequency of a variable is not observed.
- All date values will be presented as ddmmmyyyy (e.g., 29AUG2011) format. A 4-digit year is preferred for all dates.
- If applicable, all observed time values will be presented by using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds should only be reported if they were measured as part of the study.
- All tables and data listings will have the name of the program, the location, and a date stamp on the bottom of each output.

#### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xxxx), where appropriate.
- Population sizes shown with summary statistics are the samples sizes (n) of subjects with non-missing values.
- All population summaries for categorical variables will include all categories that were planned and for which the subjects may have had a response. Percentages corresponding to null categories (cells) will be suppressed; however counts and percentages of missing values may be needed.

Protocol: HZNP-ACT-302 


• All population summaries for continuous variables will include: N, mean, SD, minimum, and maximum. Other summaries (e.g., number missing, geometric mean, median, quartiles, 95% CIs, and coefficient of variation (CV) or % CV) may be used as appropriate.

- All percentages are rounded and reported to a single decimal point (xx.x %). A percentage of 100% will be reported as 100%.
- Population summaries that include P-values will report the P-value to 4 decimal places with a leading zero (0.0001). All P-values reported on default output from statistical software (i.e., SAS<sup>®</sup> Software) may be reported at the default level of precision. P-values <0.0001 should be reported as <0.0001 not 0.0000.




